CLINICAL TRIAL: NCT00666822
Title: Adherence to Endocrine Therapy in Women With Breast Cancer in Clinical Practice Settings
Brief Title: Compliance to a Hormone Therapy Regimen in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE6107; P30CA043703 (NIH); CASE6107 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2008-04-24; First posted 2008-04-25 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: compliance monitoring — To examine the relationship between adherence to endocrine therapy and variables from the Health Belief Model (i.e., perceived risk, barriers to and benefits of adherence, and cues to action such as physician recommendation) as well as measures of patient's perceptions of patient- and family-centered care in women with estrogen receptor-positive stage I-IIIA breast cancer.
Other: medical chart review — Patient's medical records are reviewed for information about the time since diagnosis, tumor characteristics, treatment, and comorbidity.
Other: questionnaire administration — Patients complete a 15 minute questionnaire on-line or by mail comprising questions of demographic and medical variables (i.e., age, race/ethnicity, marital and educational status, and medication side effects) as well as health beliefs and selected aspects of patient- and family-centered care. Data collected from the questionnaire will be stored in an Excel database.

SUMMARY:
RATIONALE: Understanding how well patients comply with their treatment regimen may help doctors plan the best treatment and ongoing care.

PURPOSE: This clinical trial is studying whether patients comply with their hormone therapy regimen in women with estrogen receptor-positive stage I, stage II, or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To examine the relationship between adherence to endocrine therapy and variables from the Health Belief Model (i.e., perceived risk, barriers to and benefits of adherence, and cues to action such as physician recommendation) as well as measures of patient's perceptions of patient- and family-centered care in women with estrogen receptor-positive stage I-IIIA breast cancer.

OUTLINE: Patients complete a 15 minute questionnaire on-line or by mail comprising questions of demographic and medical variables (i.e., age, race/ethnicity, marital and educational status, and medication side effects) as well as health beliefs and selected aspects of patient- and family-centered care. Data collected from the questionnaire will be stored in an Excel database.

Patient's medical records are reviewed for information about the time since diagnosis, tumor characteristics, treatment, and comorbidity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Women diagnosed with breast cancer

  * Stage I-IIIA disease
* Estrogen receptor (ER)-positive disease
* Must have begun prescribed hormonal therapy between December 2000 and December 2002
* No prior history of breast cancer

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Able to read and understand English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior breast surgery, axillary surgery, and radiotherapy to the breast or chest wall allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adherence to endocrine therapy | at 5 yrs
Effects of categorical predictors of compliance | at 5 yrs
Comparison of the means of each continuous predictor between compliers and non-compliers | at 5 yrs
Effects of continuous and categorical variables on compliance, controlling for other factors including age at diagnosis, race, education, and type of surgery | 5 yrs

SECONDARY OUTCOMES:
Time to discontinuation of tamoxifen as a time-to-event outcome | 5 yrs
Univariate and multivariate associations of covariates with risk of noncompliance | 5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Lois C. Friedman, PhD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States